CLINICAL TRIAL: NCT02003573
Title: An Open Label, Phase I, Dose Escalation Trial to Investigate the Maximum Tolerated Dose, Safety, Pharmacokinetics, and Efficacy of Volasertib in Combination With Decitabine in Patients >= 65 Years With Acute Myeloid Leukemia
Brief Title: Volasertib + Decitabine in Patients With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1230.30; 2013-001752-36 (EudraCT Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute

ARMS (1):
- volasertib + decitabine (Experimental): dose escalation and MTD (Maximum Tolerated Dose) Extension (Note: Decitabine is a Backbone Treatment and Volasertib is Investigational Medicinal Product (IMP))
  Interventions: Drug: decitabine iv; Drug: volasertib iv infusion

INTERVENTIONS:
Drug: decitabine iv — decitabine iv fixed dose
Drug: volasertib iv infusion — volasertib iv infusion (Body Surface Area (BSA) based dosing)

SUMMARY:
Dose Escalation (MTD Finding) Phase: To investigate the maximum tolerated dose (MTD), safety and pharmacokinetics of different volasertib administration schedules in combination with decitabine in previously untreated AML patients >= 65 years of age who are considered ineligible for standard intensive therapy, or patients with relapsed or refractory AML regardless of prior treatment status.

MTD Extension Phase: To collect additional data on safety, efficacy and pharmacokinetics of volasertib in combination with decitabine in previously untreated patients with AML >= 65 years of age and considered ineligible for standard intensive therapy.

ELIGIBILITY:
Inclusion criteria:

1. Dose Escalation Phase: patients with previously untreated AML, relapsed or refractory AML regardless of prior treatment status.
2. MTD Extension Phase: previously untreated AML (prior treatment for Myelodysplastic Syndrome(MDS) is allowed).
3. Age >= 65 years.
4. Previously untreated patients must be ineligible for receiving standard intensive therapy at the time of enrolment, in the opinion of the investigator and based on documented medical reasons.
5. Histologically or cytologically confirmed AML (except for APL, FAB (French-American-British)subtype M3) according to the World Health Organisation classification.
6. Eastern co-operative oncology group (ECOG) performance score =< 1 at screening.
7. Signed and dated written informed consent by start date of Screening Visit in accordance with Good Clinical Practice and local legislation.

Exclusion criteria:

1. MTD Extension Phase: Prior chemotherapy for AML (except for hydroxyurea). Patients can receive treatment with hydroxyurea in order to reduce high White Blood Cells count for no more than 28 days (cumulative); discontinuation of hydroxyurea at least one day prior to the study treatment is required. Please note that any prior therapy for MDS is allowed.
2. Acute promyelocytic leukemia (APL, FAB subtype M3), according to World Health Organisation classification.
3. Hypersensitivity to the trial drugs.
4. Other malignancy currently requiring active therapy (except for hormonal/anti-hormonal treatment, e.g. in prostate or breast cancer).
5. Known clinical central nervous system (CNS) symptoms deemed by the investigator to be related to leukemic CNS involvement.
6. QTcF (QT interval corrected for heart rate by the Fridericia formula) > 470 ms, calculated as the mean value of the triplicates taken at least 2 minutes apart at baseline or QTcF prolongation deemed clinically relevant by the investigator.
7. Baseline Left Ventricular Ejection Fraction of < 45% or below the lower limit of institutional normal range.
8. Aspartate amino transferase (AST) or alanine amino transferase (ALT) > 2.5 x the upper limit of normal (ULN). Patients with elevated liver enzyme(s) due to leukemic involvement are allowed up to = 5 x the ULN.
9. Total bilirubin > 1.5 x ULN. For patients with Gilbert's syndrome or elevation due to hepatic infiltrate, total bilirubin must be <4 x ULN.
10. Creatinine clearance (CLcr) < 30 ml/min (estimated creatinine clearance by the Cockcroft-Gault (C-G) equation.
11. Severe illness or organ dysfunction involving the kidneys, liver or other organ system, including active uncontrolled infection, which in the opinion of the investigator precludes treatment with decitabine or would interfere with the evaluation of the safety of the study treatment.
12. Presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) Classification of 3, unstable angina or poorly controlled arrhythmia as determined by the investigator. Myocardial infarction within 6 months prior to study entry.
13. Significant concurrent psychiatric disorder or social situation that according to the investigator's judgment would compromise patient's safety or compliance, interfere with consent, study participation, or interpretation of study results.
14. Patients with a systemic fungal, bacterial, viral, or other infection that is not controlled.
15. Contraindications for decitabine treatment according to the manufacturer's prescribing information provided in the Investigator Site File
16. Female patients of childbearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial and for a minimum of 6 months after completion of study treatment.
17. Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second medically acceptable method of contraception during the trial and for a minimum of 6 months after completion of study treatment.
18. Pregnant or breast feeding patients.
19. Treatment with any investigational drug within 2 weeks of administration of first study medication dose or within less than five half -lives of the investigational drug before treatment with the present trial drug, whichever is shorter, and / or persistence of toxicities of prior anti-leukemic therapies which are deemed clinically relevant.
20. Prior treatment with a Plk inhibitor such as volasertib or treatment in a clinical trial using a Plk inhibitory compound.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2016-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - Washington School of Medicine, St Louis, Missouri
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was originally planned to enter 127 patients into this trial; however, the development of volasertib was discontinued during the conduct of the study.
Groups:
- Volasertib 300 mg + Decitabine: Patients were treated according to dosing Schedule A in which decitabine (Dacogen®; solution for infusion) 20 mg/m2 was to be administered (Intravenous infusion) for the first 5 consecutive days of the treatment cycle (Day 1 to Day 5).
  Volasertib 300 mg (solution for infusion) was administered (Intravenous infusion) on Days 1 and 15 of the treatment cycle.
  The duration of a treatment cycle was 28 days. Number of treatment cycles was unlimited until the patient met criteria for stopping study medication.
- Volasertib 350 mg + Decitabine: Patients were treated according to dosing Schedule A in which decitabine (Dacogen®; solution for infusion) 20 mg/m2 was to be administered (Intravenous infusion) for the first 5 consecutive days of the treatment cycle (Day 1 to Day 5).
  Volasertib 350 mg (solution for infusion) was administered (Intravenous infusion) on Days 1 and 15 of the treatment cycle.
  The duration of a treatment cycle was 28 days. Number of treatment cycles was unlimited until the patient met criteria for stopping study medication.
- Volasertib 400 mg + Decitabine: Patients were treated according to dosing Schedule A in which decitabine (Dacogen®; solution for infusion) 20 mg/m2 was to be administered (Intravenous infusion) for the first 5 consecutive days of the treatment cycle (Day 1 to Day 5).
  Volasertib 400 mg (solution for infusion) was administered (Intravenous infusion) on Days 1 and 15 of the treatment cycle.
  The duration of a treatment cycle was 28 days. Number of treatment cycles was unlimited until the patient met criteria for stopping study medication.
Period: Overall Study
Arm/Group | Volasertib 300 mg + Decitabine | Volasertib 350 mg + Decitabine | Volasertib 400 mg + Decitabine
Started | 3 (Started are treated patients) | 4 (Started are treated patients) | 6 (Started are treated patients)
Completed | 0 | 0 | 0
Not Completed | 3 | 4 | 6
Not completed — Progressive disease | 2 | 0 | 1
Not completed — Other Adverse event | 0 | 1 | 1
Not completed — Refuse to take trial medication | 0 | 1 | 1
Not completed — Other than specified | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Treated set (TS): All entered patients received ≥1 dose of study medication and were included in the TS
Groups:
- Total: Total of all reporting groups
Arm/Group | Volasertib 300 mg + Decitabine | Volasertib 350 mg + Decitabine | Volasertib 400 mg + Decitabine | Total
Number analyzed (Participants) | 3 | 4 | 6 | 13
Age, Continuous [Median (Full Range); unit: years] | 71.0 [69 to 73] | 76.0 [73 to 84] | 69.5 [66 to 74] | 73.0 [66 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 6
  Male | 0 | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) Based on the Occurrence of Dose-limiting Toxicity (DLT) in Cycle 1
Description: The primary objective of the dose-escalation part of this study was to determine the MTD of volasertib in combination with decitabine. The MTD was to be identified based on the DLT information collected during the first treatment cycle of each dosing schedule. DLT was defined as a non-haematological drug-related toxicity of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥3.
  The MTD corresponded to the highest dose of volasertib and decitabine at which the incidence of DLT was ≤17% (i.e. 1/6 patients) during Cycle 1.
Time Frame: 4 weeks
Population: TS. One patient treated with volasertib 350 mg + decitabine had to be excluded because they did not receive all planned doses of volasertib and could therefore not be included in the calculation of MTD. Thus overall 12 patients were analysed instead of 13 patients.
Measure: Number; unit: Milligram (mg)
Groups:
- Volasertib + Decitabine: Patients were treated according to dosing Schedule A in which decitabine (Dacogen®; solution for infusion) was to be administered (Intravenous infusion) for the first 5 consecutive days of the treatment cycle (Day 1 to Day 5).
  Volasertib (solution for infusion) was administered (Intravenous infusion) on Days 1 and 15 of the treatment cycle. The duration of a treatment cycle was 28 days. Number of treatment cycles was unlimited until the patient met criteria for stopping study medication.
Arm/Group | Volasertib + Decitabine
Number analyzed (Participants) | 12
Milligram (mg) | 400

2. Primary Outcome: Number of Subjects With Dose Limiting Toxicities (DLT) in Cycle 1
Description: Number of subjects with Dose Limiting Toxicities (DLT) in Cycle 1 is presented
Time Frame: 4 weeks
Population: TS. One patient treated with volasertib 350 mg + decitabine had to be excluded because they did not receive all planned doses of volasertib and could therefore not be included in the calculation of MTD. Thus 3 patients were analysed instead of 4 patients for volasertib 350 mg + decitabine arm.
Measure: Number; unit: participant
Arm/Group | Volasertib 300 mg + Decitabine | Volasertib 350 mg + Decitabine | Volasertib 400 mg + Decitabine
Number analyzed (Participants) | 3 | 3 | 6
participant | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: All Adverse events with an onset after the first dose of study medication up to a period of 30 days after the last administration of study medication; up to 333 days
Groups:
- Total: Total of all arms
Arm/Group | Volasertib 300 mg + Decitabine | Volasertib 350 mg + Decitabine | Volasertib 400 mg + Decitabine | Total
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 13/13
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 6/6 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 300 mg + Decitabine (N=3) | Volasertib 350 mg + Decitabine (N=4) | Volasertib 400 mg + Decitabine (N=6) | Total (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 8
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3 | 2 | 6
Pneumonia fungal (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Volasertib 300 mg + Decitabine (N=3) | Volasertib 350 mg + Decitabine (N=4) | Volasertib 400 mg + Decitabine (N=6) | Total (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 2
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Oral mucosa haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Asthenia (General disorders) | 0 | 2 | 1 | 3
Chest pain (General disorders) | 0 | 1 | 1 | 2
Chills (General disorders) | 1 | 0 | 1 | 2
Face oedema (General disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 1 | 3
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 1
Oedema (General disorders) | 1 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 0 | 0 | 2
Pain (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 2
Anal infection (Infections and infestations) | 0 | 0 | 1 | 1
Bacteraemia (Infections and infestations) | 2 | 0 | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1
Urinary casts present (Investigations) | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 3 | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 1 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 1 | 2
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 2 | 3

LIMITATIONS AND CAVEATS:
This study was prematurely discontinued following the decision by the sponsor to discontinue the development of volasertib.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.